CLINICAL TRIAL: NCT03208868
Title: Leucine Enriched Essential Amino Acid Mixture to Reverse Muscle Loss in Cirrhosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-916
Record Dates: First submitted 2017-04-12; First posted 2017-07-06 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leucine enriched essential amino acid (Active Comparator): Patients with cirrhosis that are given a leucine enriched essential amino acid (EEA/LEU) supplement.
  Interventions: Dietary Supplement: Leucine enriched essential amino acid (EEA/LEU)
- Balanced amino acid supplement (Active Comparator): Patients with cirrhosis that are given a balanced amino acid (BAA) supplement.
  Interventions: Dietary Supplement: Balanced amino acid supplement (BAA)

INTERVENTIONS:
Dietary Supplement: Leucine enriched essential amino acid (EEA/LEU) — Patient with cirrhosis will be randomized to either take a Leucine enriched essential amino acid or a balanced amino acid supplement.
  Arms: Leucine enriched essential amino acid
Dietary Supplement: Balanced amino acid supplement (BAA) — Patient with cirrhosis will be randomized to either take a Leucine enriched essential amino acid or a balanced amino acid supplement.
  Arms: Balanced amino acid supplement

SUMMARY:
Loss of skeletal muscle mass or sarcopenia is the most common and potentially reversible complication in cirrhosis that increases morbidity and mortality before, during and after liver transplantation. No proven treatments exist for the prevention or reversal of sarcopenia in cirrhosis, primarily because the mechanisms responsible for this are unknown. Based on compelling preliminary studies and those of the co investigator, investigators hypothesize that the mechanism of reduced skeletal muscle mass in cirrhosis is due to a myostatin mediated impaired mTOR (mechanistic target of rapamycin) signaling resulting in reduced protein synthesis and increased autophagy. Investigators further postulate that leucine, a direct stimulant of mTOR, will reverse the impaired mTOR phosphorylation in the skeletal muscle of cirrhotics. The consequent increase in protein synthesis reduced autophagy will result in an increase in skeletal muscle mass. Investigators will test these hypotheses by quantifying the response to acute and long term (3 month) administration of leucine enriched essential amino acid (EAA/LEU) compared with an isonitrogenous isocaloric non-essential balanced amino acid mixture (does not stimulate protein synthesis) in cirrhotic patients. Fractional protein synthesis rate (FSR) in skeletal muscle, responses of the molecular regulatory pathways of skeletal muscle protein synthesis, and autophagy flux will be quantified in the acute and long term protocols. Tracer studies using L-[D5]-phenylalanine (Phe) as a primed constant infusion (prime 2µmol.kg-1.hr-1; constant 0.05 µmol.kg-1.hr-1) with and L [ring-D2] tyrosine, forearm plethysmography, and sequential skeletal muscle biopsies (total of 3 per study subject) will be used to quantify these outcomes. Anthropometric, clinical and body composition measures will be additional outcome measures for the long term intervention. Expression of regulatory signaling proteins, myostatin, IGF-1 (insulin like growth factor) , phospho-Akt, phospho-AMPK (activated protein kinase), phospho-mTOR and phospho-p70s6k will be quantified by Western immunoblots. Autophagy flux will be measured by quantifying expression of the autophagosome proteins.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients:
* Cirrhosis diagnosed by liver biopsy and/or clinical, biochemical and imaging evidence of cirrhosis.
* Abstinence from alcohol and/or other recreational drugs for at least 6 months
* Child's Pugh score 5-9 (inclusive).

Exclusion

* Cirrhotic patients:
* Child's score >9
* Pedal edema above the ankle
* Presence of concurrent illnesses (renal, cardiac, pulmonary, cerebrovascular, malignancy) or medication (anabolic steroids, corticosteroids) intake that affect skeletal muscle mass.
* Diabetes mellitus
* Active gastrointestinal bleeding
* Sepsis, encephalopathy
* Renal failure
* Hepatocellular carcinoma outside of Milan criteria
* Unwilling to sign informed consent or follow research procedures
* Does not meet inclusion criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-08-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare Fractional Synthesis Rate | Baseline to 90 days
  To test whether fractional synthesis of skeletal muscle proteins changes from baseline to 90 days with the administration of BAA or EAA/LEU. Fractional synthesis rate (FSR) of mixed muscle proteins will be calculated from the incorporation rate of the L- [ring D5] phenylalanine into the proteins and the free tissue phenylalanine enrichments using precursor product model: FSR= (∆Ep/t)/(∆Ec) x60x100 and expressed as %/hour. ΔEp is the increment in myofibrillar protein-bound L- [ring D5] phenylalanine enrichment, t is the time between the muscle biopsies. ∆Ec is the L- [ring D5] phenylalanine enrichments in the free intracellular pool in the muscle biopsies.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States